CLINICAL TRIAL: NCT00401076
Title: A One-year Open-label Study to Assess the Safety of Oral Long-term Use of SA-001 in Patients With Pancreatic Exocrine Insufficiency Caused by Chronic Pancreatitis or by Pancreatectomy
Brief Title: A Open-label Study to Assess the Safety of Oral Long-term Use of SA-001 in Pancreatic Exocrine Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Toshiaki Yamaguchi, Sr. Clinical Project Manager, Abbott
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S245.3.123
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Pancreatic Exocrine Insufficiency, Chronic Pancreatitis, Pancreatectomy
Keywords: SA-001; Pancreatic Exocrine Insufficiency; Chronic Pancreatitis; Pancreatectomy
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SA-001

INTERVENTIONS:
Drug: SA-001 — 0.25 g of SA-001 pellets/capsule, 12 capsules/day for 52 weeks

SUMMARY:
This study is to evaluate the safety of 3.0 g/day of SA-001 (to be flexibly increased or decreased with the range from 1.5 g/day to 6.0 g/day), which will orally be administered for 52 weeks to patients with pancreatic exocrine insufficiency caused by chronic pancreatitis in the non-compensatory stage or by pancreatectomy.

ELIGIBILITY:
Inclusion Criteria Subjects who complete the S245.3.122 clinical study (excluding discontinued subjects).

Exclusion Criteria Subjects who are assessed to be inappropriate for continuing long-term use of SA-001, at the discretion of the investigator or the sub-investigator, because they experienced adverse drug reactions in the S245.3.122 clinical study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety of long-term use of 3.0 g/day SA 001 (12 capsules/day), flexibly increased or decreased within the range of 1.5 g/day SA 001 (6 capsules/day) to 6.0 g/day SA-001 (24 capsules/day) | 52 weeks

SECONDARY OUTCOMES:
Efficacy data (nutritional evaluation items) of 3.0 g/day SA-001 (12 capsules/day), flexibly increased or decreased within the range of 1.5 g/day SA 001 (6 capsules/day) to 6.0 g/day SA-001 (24 capsules/day) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Yamaguchi, BS Pharm, Study Director — Abbott
Locations (17):
- Japan (17):
  - Site Reference ID/Investigator# 45211, Fukuoka
  - Site Reference ID/Investigator# 45297, Fukuoka
  - Site Reference ID/Investigator# 45220, Hiroshima
  - Site Reference ID/Investigator# 45279, Hiroshima
  - Site Reference ID/Investigator# 45223, Hokkaido
  - Site Reference ID/Investigator# 45303, Hokkaido
  - Site Reference ID/Investigator# 45091, Hyōgo
  - Site Reference ID/Investigator# 45110, Kanagawa
  - Site Reference ID/Investigator# 45213, Kanagawa
  - Site Reference ID/Investigator# 45207, Kyoto
  - Site Reference ID/Investigator# 45111, Miyagi
  - Site Reference ID/Investigator# 45282, Miyagi
  - Site Reference ID/Investigator# 45283, Nagasaki
  - Site Reference ID/Investigator# 45106, Osaka
  - Site Reference ID/Investigator# 45242, Sapporo
  - Site Reference ID/Investigator# 45281, Tokyo
  - Site Reference ID/Investigator# 45299, Yamaguchi